CLINICAL TRIAL: NCT06322797
Title: A Randomized, Controlled, Patient- and Assessor- Blinded, Exploratory Clinical Trial to Search the Stimulation Site for Repetitive Transcranial Magnetic Stimulation (rTMS) That Improves Upper Extremity Function After Stroke
Brief Title: The Safety&Efficacy of Repetitive Transcranial Magnetic Stimulation for Post-Stroke Upper Extremity Function Improvement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MinYoung Kim, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, MD, PhD, Professor of CHA university, M.D., Ph.D., Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rTMSinStroke
Record Dates: First submitted 2022-07-12; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: Stroke; Functional Magnetic Resonance Imaging; Repetitive transcranial magnetic stimulation; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMS over the M1 cortex of the injured hemisphere localized by motor action potential (Experimental): Experimental A group : rTMS was administered by trained physicians over the M1 cortex of the injured hemisphere aiming at the site that caused the largest visible twitch in the participant's thumb.
  Interventions: Device: rTMS
- rTMS over the specific site of the injured hemisphere localized by fMRI (Experimental): Experimental B group : rTMS was administered by trained physicians over the specific site which is after checking the brain site activated during finger tapping during fMRI imaging, target coordinates are set based on the 10-20 EEG system coordinate system in the taken MRI image.
  Interventions: Device: rTMS
- Sham group (Sham Comparator): Sham group: shame rTMS( sound mode) is applied over the M1 cortex of the injured hemisphere which is the site that caused the largest visible twitch in the participant's thumb when stimulation is applied
  Interventions: Device: Sham

INTERVENTIONS:
Device: rTMS — Stimulation was performed using a biphasic stimulator (ALTMS® Remed, Republic of Korea) and a 70-mm figure-eight coil. The routine stimulation procedure is described as follows. First, the resting motor threshold was measured for each patient. At the lowest stimulus output, a stimulus was applied to the M1 cortex of the uninjured hemisphere aiming at the site that caused the largest visible twitch in the participant's thumb. The resting motor threshold was defined as the intensity required to generate a motor-induced potential of > 50 uV in the contralateral abductor pollicis brevis muscle at least 5 out of 10 times with 30 s of inter-stimulus time interval.
  Stimulation was given at 100% of the resting motor threshold stimulator output: 20 Hz, 5-s train duration, 55-s inter-train interval, and a total number of stimulations of 2000 pulses per session for 20 min.
  Arms: rTMS over the M1 cortex of the injured hemisphere localized by motor action potential
Device: rTMS — Stimulation was performed using a biphasic stimulator (ALTMS® Remed, Republic of Korea) and a 70-mm figure-eight coil. The routine stimulation procedure is described as follows. After identifying the brain site that is activated during finger tapping during fMI, Stimulation was given at 100% of the resting motor threshold stimulator output: 20 Hz, 5-s train duration, 55-s inter-train interval, and a total number of stimulations of 2000 pulses per session for 20 min. the resting motor threshold was measured for each patient at target brain site.
  Arms: rTMS over the specific site of the injured hemisphere localized by fMRI
Device: Sham — In Sound Mode, no actual stimulation is applied, and 20 minutes of treatment is performed like other experimental groups.
  Arms: Sham group

SUMMARY:
A randomized, controlled, subject and rater-blind, exploratory clinical trial to evaluate the safety and efficacy of repetitive transcranial magnetic stimulation for improvement of upper extremity function after stroke.

DETAILED DESCRIPTION:
Some studies related to rTMS for the recovery of motor function (upper and lower extremity functions) after stroke are being conducted, and the clear mechanism has not been elucidated. It is known that function is restored through various neurophysiological changes.

However, there are not many studies on rTMS in the chronic stroke period, 3 months after the onset of stroke recovery, which is slow, and among them, there is no established standard for which part of the brain should be stimulated for treatment.

Recently, techniques for finding brain regions that are activated when performing a specific action through an imaging technique called fMRI (Functional Magnetic Resonance Imaging) are being used in various fields.

Based on the idea in this regard, recent studies have been conducted that the effect of rTMS treatment is better than the existing method when fMRI is used to identify the brain regions involved in the movement of the upper and lower extremities.

The purpose of this study is to evaluate the safety and efficacy on upper extremity function after stroke using fMRI and rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years of age
* Patients 3 months or more after stroke onset
* Patients with NIHSS score of 1 or more to 20 or less
* After hearing and fully understanding the detailed explanation of this clinical trial, the subject or legal representative voluntarily decides to participate and agrees in writing to abide by the precautions

Exclusion Criteria: Patients who fall under one or more of the following conditions are not eligible to participate in the study.

* Patients with systemic infectious disease at the time of participation in the clinical trial
* In the case of a person with impaired consent (MMSE less than 10 points), if not accompanied by a guardian
* Those with severe medical conditions such as unstable conditions of the cardiovascular system, digestive system, respiratory system, endocrine system, etc., who are in poor general condition
* Other cases where the researcher determines that participation in this clinical trial is not appropriate
* Those who are contraindicated in repetitive transcranial magnetic stimulation A. When metal materials (deep brain stimulation electrode, brain aneurysm clip, cardiac pacemaker, etc.) are in the body B. Uncontrolled epilepsy (epilepsy), patients with psychiatric disorders
* Pregnant, lactating women and patients with potential for pregnancy
* Patients with contraindications for imaging tests
* Those who have undergone cerebral surgery due to past or current related medical history

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Fugl-Meyer Assessment | Baseline - 1month - 3months
  The difference in the FMA (Fugl-Meyer Assessment) between the three groups at baseline, 30 days and 90 days was confirmed by comparing differences.[0~66 for each arm] (The higher values represent a better outcome.)

SECONDARY OUTCOMES:
Change of Range of motion | Baseline - 1month - 3months
  The difference in the ROM(Range of motion between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.
Change of Berg Balance Scale | Baseline - 1month - 3months
  The difference in the BBS (Berg Balance Scale) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.[0~56] (The higher values represent a better outcome.)
Change of Motor Assessment Scale | Baseline - 1month - 3months
  The difference in the MAS (Motor Assessment Scale) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.[0~54] (The higher values represent a better outcome.)
Change of Trunk Imbalance Scale | Baseline - 1month - 3months
  The difference in the TIS (Trunk Imbalance Scale) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.[0~23] (The higher values represent a better outcome.)
Change of Functional Ambulation Category | Baseline - 1month - 3months
  The difference in the FAC (Functional Ambulation Category) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.[0~5] (The higher values represent a better outcome.)
Change of Time up and go | Baseline - 1month - 3months
  The difference in the TUG (Time up and go) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences. (The lower values represent a better outcome.)
Change of Manual muscle Test | Baseline - 1month - 3months
  The difference in the MMT (Manual muscle test) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.[0~5 for each muscle] (The higher values represent a better outcome.)
Change of Action reach arm test | Baseline - 1month - 3months
  The difference in the ARAT(Action reach arm test) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.[0~57] (The higher values represent a better outcome.)
Change of Jebsen taylor hand function test | Baseline - 1month - 3months
  The difference in the Jebsen taylor hand function test between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences. (The lower values represent a better outcome.)
Change of Functional Independence Measure | Baseline - 1month - 3months
  The difference in the FIM (Functional Independence Measure) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.[0~126] (The higher values represent a better outcome.)
Change of Modified Barthel index | Baseline - 1month - 3months
  The difference in the MBI (Modified Barthel index) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.[0~100] (The higher values represent a better outcome.)
Change of National Institutes of Health Stroke Scale | Baseline - 1month - 3months
  The difference in the NIHSS (National Institutes of Health Stroke Scale) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.[0~42] (The lower values represent a better outcome.)
Change of Korean Mini Mental State Exam | Baseline - 1month - 3months
  The difference in the K-MMSE (Korean Mini Mental State Exam) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences. [0~30] (The higher values represent a better outcome.)
Change of Clinical Dementia Rating | Baseline - 1month - 3months
  The difference in the CDR(clinical dementia rating) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences. [0~5] (The lower values represent a better outcome.)
Change of Global Deterioration Scale | Baseline - 1month - 3months
  The difference in the GDS(Global Deterioration Scale) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences. [0~7] (The lower values represent a better outcome.)
Change of Geriatric Depression Scale | Baseline - 1month - 3months
  The difference in the GDSd(Geriatric Depression Scale) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences. [0~30] (The lower values represent a better outcome.)
Change of Brain imaging | Baseline - 1month - 3months
  The difference in the Brain imaging (functional brain MRI) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences. (Only in Experimental B group)
Change of Electroencephalography | Baseline - 1month - 3months
  The difference in the Electroencephalography between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences. ( Band power of the multiple brain sites based on the 10-20 EEG system [Frontal (Fp1, Fp2, F7, F3, Fz, F4, F8), Central (C3, Cz, C4),Temporal (T3,T4,T5,T6), Parietal (P3, Pz, P4), Occipital (O1, O2)] measured in the various EEG frequency bands [(Delta (1~4Hz), Theta (4~8Hz), Alpha1 (8~10Hz), Alpha2 (10~12Hz), Beta1 (12~15Hz), Beta2 (15~20Hz), Beta3 (20~30Hz), Gamma (30~45Hz)]
Change of Evoked Potential | Baseline - 1month - 3months
  The difference in the EP(Evoked Potential) Study between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.
Changes in test results of WBC(/uL), RBC(/uL), , Hct(%), PLT(/uL), Hgb(g/dL) | Baseline - 1month - 3months
  The difference in the Laboratory test WBC(/uL), RBC(/uL), , Hct(%), PLT(/uL), Hgb(g/dL) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.
Changes in test results of CRP (mg/dL), glucose (mg/dL), BUN (mg/dL), creatinine (mg/dL), total cholesterol (mg/dL) | Baseline - 1month - 3months
  The difference in the Laboratory test [CRP(mg/dL), Glucose(mg/dL), BUN(mg/dL) , Creatinine(mg/dL), Total choliesterol(mg/dL)] between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.
Changes in test results of AST(IU/L), ALT(IU/L) | Baseline - 1month - 3months
  The difference in the Laboratory test [AST(IU/L), ALT(IU/L)] between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences.
Change of Motricity index | Baseline - 1month - 3months
  The difference in the MI(Motricity index) between the three groups at baseline, 30 days, and 90 days was confirmed by comparing differences. [0~100] (The higher values represent a better outcome.)

CONTACTS AND LOCATIONS:
Overall Officials: Kim MinYoung, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- Department of Rehabilitation Medicine, CHA Bundang Medical Center, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No